CLINICAL TRIAL: NCT02747186
Title: Pilot Study: Comparison of Buffered 1% vs. Non-Buffered 2% Lidocaine Used in Dental and Oral Surgical Procedures: Clinical Outcomes Maxilla
Brief Title: Clinical Outcomes Maxilla: Buffered 1% Lidocaine vs. Non-buffered 2% Lidocaine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 16-0068b
Record Dates: First submitted 2016-04-19; First posted 2016-04-21 (Estimated); Results first posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-10

CONDITIONS: Anesthesia
Keywords: lidocaine, jaw
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Buffered 1% lidocaine (Active Comparator): In week One each subject would receive the anesthetic, 5cc, to block the Posterior alveolar, Anterior alveolar, Palatal nerves.Maxillary molar and canine tested for pulpal anesthesia.
  At least a week later, injections for the maxillary field block would involve the alternate local anesthetic combination. Maxillary molar and canine tested for pulpal anesthesia.
  Interventions: Drug: Lidocaine
- Non-Buffered lidocaine (Active Comparator): In week One each subject would receive the anesthetic, 5cc, to block the Posterior alveolar, Anterior alveolar, Palatal nerves. Maxillary molar and canine tested for pulpal anesthesia.
  At least a week later, injections for the maxillary field block would involve the alternate local anesthetic combination. Maxillary molar and canine tested for pulpal anesthesia.
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — Intraoral maxillary field block
  Other Names: xylocaine

SUMMARY:
Anecdotal data suggest that the buffered form of the local anesthetic is more potent at equal dosages, and a lower dosage of the buffered drug might be used with an effect equal to higher dosage not buffered. Clinical data are needed to confirm these anecdotal data. No published data exist comparing buffered local anesthetics at lower drug concentrations to current dosages commonly used in dental and oral surgical procedures

DETAILED DESCRIPTION:
Specific Aims:

Compare clinical depths of pulpal anesthesia for maxillary molar and canine teeth at 30min intervals post injection after maxillary field block anesthesia with buffered 1% lidocaine with 1/100,000 epinephrine as compared to non-buffered 2% lidocaine with 1/100,000 epinephrine.

Hypotheses:

No differences exist in anesthetic depth for pulpal anesthesia after intraoral injection for maxillary field block anesthesia between buffered 1% lidocaine with 1/100,000 epinephrine as compared to non-buffered 2% lidocaine with 1/100,000 epinephrine.

Study Time Frame: 6 months: Month One Recruit 24 volunteers as subjects, Prepare case-books. Months Two-Three Clinical Study. Months Four-Five Analyze Lab data. Month Six Prepare Abstracts, Papers Methods: Blinded, Randomized Clinical Design, Recruit subjects with Institutional Review Board approved consent at University of North Carolina. Subjects will serve as their own controls in a cross-over AB/BA study design which is uniform within sequences, uniform within periods, and balanced. Randomized subjects to be injected orally for maxillary field block (Posterior alveolar, Anterior alveolar, Palatal sensory nerves) alternatively with 4cc of buffered 1% lidocaine with 1/100,000 epinephrine and 4cc non-buffered of 2% lidocaine with 1/100,000 epinephrine.

Assessment: pre, and post-anesthetic administration for pulpal anesthesia with cold, electronic pulp test at maxillary molar and canine at 30 minute intervals.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists Risk Classification I Willingness to participate in two sessions

Exclusion Criteria:

* Allergy to lidocaine class of anesthetic drugs Local anesthetic drug use in past week Current symptoms teeth or oral mucosa

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-05; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond P White, Jr., DDS, PhD, Principal Investigator — UNC Department Oral and Maxillofacial Surgery
Locations (1):
- University of North Carolina School of Dentistry, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
No Plans

RESULTS

PARTICIPANT FLOW:
Groups:
- Buffered 1% Lidocaine, Then Non-Buffered 2% Lidocaine; Non-Buffered 2% Lidocaine, Then Buffered 1% Lidocaine: At each treatment visit, participants were injected orally for maxillary field block (Posterior alveolar, Anterior alveolar, Palatal nerves).
Period: First Intervention
Arm/Group | Buffered 1% Lidocaine, Then Non-Buffered 2% Lidocaine | Non-Buffered 2% Lidocaine, Then Buffered 1% Lidocaine
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Washout (1 Week)
Arm/Group | Buffered 1% Lidocaine, Then Non-Buffered 2% Lidocaine | Non-Buffered 2% Lidocaine, Then Buffered 1% Lidocaine
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Buffered 1% Lidocaine, Then Non-Buffered 2% Lidocaine | Non-Buffered 2% Lidocaine, Then Buffered 1% Lidocaine
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants who were randomized to receive either Buffered 1% Lidocaine or Non-Buffered 2% Lidocaine
Arm/Group | All Study Participants
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 24 [21 to 26]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Mean Time to Pulpal Response After Maxillary Molar Anesthesia
Description: Subjects' maxillary molar teeth will be tested before anesthetic and every 30 minutes with cold and electronic pulp test for presence of anesthesia as reported by subjects yes or no.
Time Frame: Every 30 minutes up to 120 minutes Total
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Buffered 1% Lidocaine: All subjects who received Buffered 1% Lidocaine.
- Non-Buffered 2% Lidocaine: All subjects who received Non-Buffered 2% Lidocaine.
Arm/Group | Buffered 1% Lidocaine | Non-Buffered 2% Lidocaine
Number analyzed (Participants) | 24 | 24
minutes | 98.8 (30.6) | 84.5 (27)

2. Primary Outcome: Mean Time to Pulpal Response After Maxillary Canine Anesthesia
Description: as for outcome 1
Time Frame: Every 30 minute up to 120 minutes total
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Buffered 1% Lidocaine | Non-Buffered 2% Lidocaine
Number analyzed (Participants) | 24 | 24
minutes | 77.1 (30.8) | 70.9 (35.3)

ADVERSE EVENTS:
Time Frame: Adverse events collected for 24 hours following each of the injections administered during both treatment interventions
Groups:
- Buffered 1% Lidocaine; Non-Buffered 2% Lidocaine: In week One, each subject would receive the anesthetic, 5cc, to block the Posterior alveolar, Anterior alveolar, Palatal nerves. Maxillary molar and canine tested for pulpal anesthesia. At least a week later, injections for the maxillary field block would involve the alternate local anesthetic combination. Maxillary molar and canine tested for pulpal anesthesia.
Arm/Group | Buffered 1% Lidocaine | Non-Buffered 2% Lidocaine
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-21): https://cdn.clinicaltrials.gov/large-docs/86/NCT02747186/Prot_SAP_000.pdf